CLINICAL TRIAL: NCT06025448
Title: From Cuff Arthropathy to Reverse Shoulder Arthroplasty - a Multicentre Randomized Control Trial (CARS 2: Is MIO-RSA Noninferior to BIO-RSA When it Comes to Mechanical Implant Stability Measured With CT-based Motion Analysis (CTMA)?).
Brief Title: Is MIO-RSA Noninferior to BIO-RSA When it Comes to Mechanical Implant Stability?
Acronym: CARS-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARS-2
Record Dates: First submitted 2023-06-28; First posted 2023-09-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Arthroplasty Complications; Shoulder Osteoarthritis
Keywords: Reverse shoulder arthroplasty; BIO-RSA; MIO-RSA; Bony lateralization; Metallic lateralization; Orthopedic Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and health personnel examining the participants will be blinded. It will not be possible to blind the surgeons due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIO-RSA (Active Comparator)
  Interventions: Procedure: BIO-RSA
- MIO-RSA (Experimental)
  Interventions: Procedure: MIO-RSA

INTERVENTIONS:
Procedure: BIO-RSA — Patients will have a reversed shoulder arthroplasty with lateralization of the joint centre using bony lateralization (BIO-RSA).
  Arms: BIO-RSA
Procedure: MIO-RSA — Patients will have a reversed shoulder arthroplasty with lateralization of the joint centre using metallic lateralization (MIO-RSA).
  Arms: MIO-RSA

SUMMARY:
This clinical trial will investigate whether metallic lateralization in reverse shoulder arthroplasty is as stable as bony lateralization during the first two postsurgical years, measured with CT-based motion analysis (CTMA).

DETAILED DESCRIPTION:
Lateralization of reverse shoulder arthroplasties may reduce the risk for complications such as limited range of motion (ROM), and scapular notching, where the lower part of the scapular neck becomes eroded due to impingement against the humeral component. There's several ways to lateralize the glenoid component, a bone transplant placed underneath the glenoid component (Bony Increased Offset Reversed Shoulder Arthroplasty: BIO-RSA) has been used for some time. Recently glenoid components with metallic lateralization of the joint centre (Metal-Increased Offset Reversed Shoulder Arthroplasty: MIO-RSA) have been introduced, but there is not much comparative literature on metal vs. bony lateralization.

Patients with osteoarthritis and medialization of the glenoid articular surface, who willing to participate in a study will be randomized to receive either MIO-RSA or a BIO-RSA. CT-based motion analysis (CTMA) will be used to measure the 3-dimensional migration pattern of the glenoid components to assess the stability of the prostheses up to two years after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for primary RSA due to OA, massive RC tear, failed RC repair or post-instability osteoarthritis
* massive glenoid medialization
* Able to read or write Norwegian

Exclusion Criteria:

* Severe osteoporosis
* Osteonecrosis of the humeral head
* Dementia
* Poor deltoid function
* Revision surgery
* ASA IV
* Suspected chronic infection
* Acute fracture

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2033-03-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Migration of glenoid component from baseline until 24 months | At baseline and 3, 6, 12 and 24 months postoperatively. 24 months will be the primary outcome.
  CT-based motion analysis (CTMA) will be used to measure the 3-dimensional migration pattern of the glenoid components to assess the stability of the prostheses up to two years after implantation.
  The motion analysis includes measurement of translation along three orthogonal axes and rotations around two orthogonal axes. CTMA is a marker-free motion analysis, and the images are obtained on a standard CT-machine. Analysis and computation of motion data are performed using proprietary software at Sectra AB (collaborating partner)
  CTMA is a relative new method to measure implant migration. The precision of the measurements is 0.08-0.15 mm for translation and 0.23-0.54º for rotation, therefore, CTMA is capable of measuring very small movements of the implant relative to the surrounding bone.

SECONDARY OUTCOMES:
Change in WOOS Index | Before randomization, 3, 12 and 24 months postoperatively.
  The Western Ontario Osteoarthritis of the Shoulder (WOOS) index is a patient-reported, disease-specific questionnaire for the measurement of the quality-of-life in patients with osteoarthritis.
  There are 19 questions divided into four domains: Physical symptoms, sports and work, lifestyle and emotions. Each question is answered on a visual analogue scale ranging from 0 to 100. The overall score ranges from 0 to 1900, with 1900 being the worst. For ease of interpretation, the scores are often converted to a percentage of the maximum score.
Change in Constant-Murley Score | Before randomization, 3, 12 and 24 months postoperatively.
  The CMS is a multi-item functional scale assessing pain, ADL, ROM and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively. The test is divided into subjective and objective components. Two subjective: pain and activities of daily living (ADL) and two objective: range of motion (ROM) and strength. The subjective components can receive up to 35 points and the objective 65.
  Pain and ADL are answered by the patient; ROM and strength require a physical evaluation and are answered by the orthopaedic surgeon or the physiotherapist.
Change in EuroQol-5 | Before randomization, 3, 12 and 24 months postoperatively.
  he widely used EuroQol-5 (EQ-5D-5L) will be used to measure health-related quality of life.
  The EQ5D-5L consists of two parts: A descriptive system (Mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and the EQ-VAS that record patients self-rated health on a visual analog scale that range from 0 -100, higher levels indicate better self-rated health.
  The descriptive system can be converted to a single summary index number where lower levels indicate poorer health related quality of life.
Change in range of motion | Before randomization, 3, 12 and 24 months postoperatively.
  The patient's active and passive range of motion (ROM) in the affected shoulder will be measured by an experienced physiotherapist with a long-legged goniometer. The directions measured will be flexion, abduction, external rotation and internal rotation, measured in degrees and/or physical landmarks.
Change in Subjective Shoulder Value | Before randomization, 3, 12 and 24 months postoperatively.
  The SSV score is defined as the subjective evaluation by the patient of shoulder function, expressed as a percentage of a normal shoulder. This score ranges from 0 to 100%.
Anchor Question 1 | Before randomization, 3, 12 and 24 months postoperatively.
  This anchor question is asked to help determine Patient Acceptable Symptom State (PASS).
  "Considering all daily activities that involves your operated shoulder, your level of pain and degree of function, how satisfied are you with the condition of your shoulder is right now?" Alternatives: Satisfied/somewhat satisfied/Neither satisfied or unsatisfied/somewhat unsatisfied/Unsatisfied
Anchor Question 2 | 3, 12 and 24 months postoperatively
  This anchor question is asked to help determine Minimal Important Difference (MID) and Substantial Clinical Benefit (SCB).
  "Think of all the ways your operated shoulder has affected you the last week. Since your surgery, has there been any change in the condition of your shoulder that you would consider important or meaningful to you?" Alternatives: Much better/moderately better/a bit better/no change/a bit worse/moderately worse/Much worse

CONTACTS AND LOCATIONS:
Overall Officials: Sigbjørn Dimmen, Prof., Principal Investigator — University of Oslo; Kjersti Kaul Jenssen, PhD, Principal Investigator — Lovisenberg Diaconal Hospital; Christian Owesen, PhD, Study Director — Lovisenberg Diaconal Hospital
Locations (1):
- Lovisenberg Diaconal Hospital, Oslo, Norway